CLINICAL TRIAL: NCT03180775
Title: Effects of Dietary Amino Acids on Serum and Macrophage Atherogenicity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Prof. Tony hayek MD, Director, Department of Internal Medicine E, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0566-16-RMB CTIL
Record Dates: First submitted 2017-05-25; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Atherosclerosis; Diet Modification; Serum; Disease
Keywords: Amino acids; Macrophage atherogenicity; Triglycerides; Cholesterol; Lipoproteins
MeSH Terms: conditions — Atherosclerosis; Disease | interventions — Cellulose; Glycine; Alanine; Leucine; Isoleucine; Valine; Cysteine; Arginine; Methionine; Glutamic Acid; Glutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Control (Sham Comparator): Other: Cellulose (control): cellulose, water soluble powder, 2 g in one daily dose, during 30 days
  Interventions: Other: Cellulose (control)
- Glycine (Trade name: Glycine) (Experimental): Dietary Supplement: Glycine, water soluble powder, 7.8 g daily in one dose, during 30 days.
  Interventions: Dietary Supplement: Glycine
- Alanine (Trade name: L-Alanine) (Experimental): Dietary Supplement: Alanine, water soluble powder, 8.5 g daily in one dose, during 30 days.
  Interventions: Dietary Supplement: Alanine
- Leucine (Trade name: L-Leucine) (Experimental): Dietary Supplement: Leucine, water soluble powder, 14 g daily in one dose, during 30 days.
  Interventions: Dietary Supplement: Leucine
- Isoleucine (Trade name: L-Isoleucine) (Experimental): Dietary Supplement: Isoleucine, water soluble powder, 8.2 g daily in one dose, during 30 days.
  Interventions: Dietary Supplement: Isoleucine
- Valine (Trade name: L-Valine) (Experimental): Dietary Supplement: Valine, water soluble powder, 9 g daily in one dose, during 30 days.
  Interventions: Dietary Supplement: Valine
- Cysteine (Trade name: L-Cysteine) (Experimental): Dietary Supplement: Cysteine, water soluble powder, 2.2 g daily in one dose, during 30 days.
  Interventions: Dietary Supplement: Cysteine
- Arginine (Trade name: L-Arginine) (Experimental): Dietary Supplement: Arginine, water soluble powder, 10 g daily in one dose, during 30 days.
  Interventions: Dietary Supplement: Arginine
- Methionine (Trade name: DL-Methionine) (Experimental): Dietary Supplement: Methionine, water soluble powder, 4 g daily in one dose, during 30 days.
  Interventions: Dietary Supplement: Methionine
- Glutamate (Trade name: L-Glutamic acid) (Experimental): Dietary Supplement: Glutamate, water soluble powder, 33 g daily in one dose, during 30 days.
  Interventions: Dietary Supplement: Glutamate
- Glutamine (Trade name: L-Glutamine) (Experimental): Dietary Supplement: Glutamine, water soluble powder, 30 g daily in one dose, during 30 days.
  Interventions: Dietary Supplement: Glutamine

INTERVENTIONS:
Other: Cellulose (control) — Cellulose (a vegetal product, in powder form, used as dietary fiber, that is not digested or absorbed in the intestines), will be supplemented in the form of water soluble powder.
  Arms: Control
Dietary Supplement: Glycine — Amino acids are the building blocks of proteins, they are essential organic compounds in the normal diet, and are also individually administered as nutritional supplements. Glycine will be supplied in the form of water soluble powder (the commercial form), for one daily dose. The corresponding amino acid doses were established based on the highest intakes at the 99th percentile in adult men (Institute of Medicine. 2005. Dietary Reference Intakes for Energy, Carbohydrate, Fiber, Fat, Fatty Acids, Cholesterol, Protein, and Amino Acids. Washington, D.C.: The National Academies Press. doi.org/10.17226/10490).
  Other Names: Trade name: Glycine (Manufacturer Fagron Inc)
  Arms: Glycine (Trade name: Glycine)
Dietary Supplement: Alanine — Amino acids are the building blocks of proteins, they are essential organic compounds in the normal diet, and are also individually administered as nutritional supplements. Alanine will be supplied in the form of water soluble powder (the commercial form), for one daily dose. The corresponding amino acid doses were established based on the highest intakes at the 99th percentile in adult men (Institute of Medicine. 2005. Dietary Reference Intakes for Energy, Carbohydrate, Fiber, Fat, Fatty Acids, Cholesterol, Protein, and Amino Acids. Washington, D.C.: The National Academies Press. doi.org/10.17226/10490).
  Other Names: Trade name: L-Alanine (Manufacturer Fagron Inc)
  Arms: Alanine (Trade name: L-Alanine)
Dietary Supplement: Leucine — Amino acids are the building blocks of proteins, they are essential organic compounds in the normal diet, and are also individually administered as nutritional supplements. Leucine will be supplied in the form of water soluble powder (the commercial form), for one daily dose. The corresponding amino acid doses were established based on the highest intakes at the 99th percentile in adult men (Institute of Medicine. 2005. Dietary Reference Intakes for Energy, Carbohydrate, Fiber, Fat, Fatty Acids, Cholesterol, Protein, and Amino Acids. Washington, D.C.: The National Academies Press. doi.org/10.17226/10490).
  Other Names: Trade name: L-Leucine (Manufacturer Fagron Inc)
  Arms: Leucine (Trade name: L-Leucine)
Dietary Supplement: Isoleucine — Amino acids are the building blocks of proteins, they are essential organic compounds in the normal diet, and are also individually administered as nutritional supplements. Isoleucine will be supplied in the form of water soluble powder (the commercial form), for one daily dose. The corresponding amino acid doses were established based on the highest intakes at the 99th percentile in adult men (Institute of Medicine. 2005. Dietary Reference Intakes for Energy, Carbohydrate, Fiber, Fat, Fatty Acids, Cholesterol, Protein, and Amino Acids. Washington, D.C.: The National Academies Press. doi.org/10.17226/10490).
  Other Names: Trade name: L-Isoleucine (Manufacturer Fagron Inc)
  Arms: Isoleucine (Trade name: L-Isoleucine)
Dietary Supplement: Valine — Amino acids are the building blocks of proteins, they are essential organic compounds in the normal diet, and are also individually administered as nutritional supplements. Valine will be supplied in the form of water soluble powder (the commercial form), for one daily dose. The corresponding amino acid doses were established based on the highest intakes at the 99th percentile in adult men (Institute of Medicine. 2005. Dietary Reference Intakes for Energy, Carbohydrate, Fiber, Fat, Fatty Acids, Cholesterol, Protein, and Amino Acids. Washington, D.C.: The National Academies Press. doi.org/10.17226/10490).
  Other Names: Trade name: L-Valine (Manufacturer Fagron Inc)
  Arms: Valine (Trade name: L-Valine)
Dietary Supplement: Cysteine — Amino acids are the building blocks of proteins, they are essential organic compounds in the normal diet, and are also individually administered as nutritional supplements. Cysteine will be supplied in the form of water soluble powder (the commercial form), for one daily dose. The corresponding amino acid doses were established based on the highest intakes at the 99th percentile in adult men (Institute of Medicine. 2005. Dietary Reference Intakes for Energy, Carbohydrate, Fiber, Fat, Fatty Acids, Cholesterol, Protein, and Amino Acids. Washington, D.C.: The National Academies Press. doi.org/10.17226/10490).
  Other Names: Trade name: L-Cysteine (Manufacturer Fagron Inc)
  Arms: Cysteine (Trade name: L-Cysteine)
Dietary Supplement: Arginine — Amino acids are the building blocks of proteins, they are essential organic compounds in the normal diet, and are also individually administered as nutritional supplements. Arginine will be supplied in the form of water soluble powder (the commercial form), for one daily dose. The corresponding amino acid doses were established based on the highest intakes at the 99th percentile in adult men (Institute of Medicine. 2005. Dietary Reference Intakes for Energy, Carbohydrate, Fiber, Fat, Fatty Acids, Cholesterol, Protein, and Amino Acids. Washington, D.C.: The National Academies Press. doi.org/10.17226/10490).
  Other Names: Trade name: L-Arginine (Manufacturer Fagron Inc)
  Arms: Arginine (Trade name: L-Arginine)
Dietary Supplement: Methionine — Amino acids are the building blocks of proteins, they are essential organic compounds in the normal diet, and are also individually administered as nutritional supplements. Methionine will be supplied in the form of water soluble powder (the commercial form), for one daily dose. The corresponding amino acid doses were established based on the highest intakes at the 99th percentile in adult men (Institute of Medicine. 2005. Dietary Reference Intakes for Energy, Carbohydrate, Fiber, Fat, Fatty Acids, Cholesterol, Protein, and Amino Acids. Washington, D.C.: The National Academies Press. doi.org/10.17226/10490).
  Other Names: Trade name: DL-Methionine (Manufacturer Fagron Inc)
  Arms: Methionine (Trade name: DL-Methionine)
Dietary Supplement: Glutamate — Amino acids are the building blocks of proteins, they are essential organic compounds in the normal diet, and are also individually administered as nutritional supplements. Glutamate will be supplied in the form of water soluble powder (the commercial form), for one daily dose. The corresponding amino acid doses were established based on the highest intakes at the 99th percentile in adult men (Institute of Medicine. 2005. Dietary Reference Intakes for Energy, Carbohydrate, Fiber, Fat, Fatty Acids, Cholesterol, Protein, and Amino Acids. Washington, D.C.: The National Academies Press. doi.org/10.17226/10490).
  Other Names: Trade name: L-Glutamic acid (Manufacturer Fagron Inc)
  Arms: Glutamate (Trade name: L-Glutamic acid)
Dietary Supplement: Glutamine — Amino acids are the building blocks of proteins, they are essential organic compounds in the normal diet, and are also individually administered as nutritional supplements. Glutamine will be supplied in the form of water soluble powder (the commercial form), for one daily dose. The corresponding amino acid doses were established based on the highest intakes at the 99th percentile in adult men (Institute of Medicine. 2005. Dietary Reference Intakes for Energy, Carbohydrate, Fiber, Fat, Fatty Acids, Cholesterol, Protein, and Amino Acids. Washington, D.C.: The National Academies Press. doi.org/10.17226/10490).
  Other Names: Trade name: L-Glutamine (Manufacturer Fagron Inc)
  Arms: Glutamine (Trade name: L-Glutamine)

SUMMARY:
Recently, the investigators have been screening for anti-atherogenic or pro-atherogenic amino acids (AAs) in the macrophage model system to better understand their role in atherogenesis. The findings so far suggest that specific AAs induce selective anti-atherogenic effects (glycine, alanine, leucine and cysteine) or pro-atherogenic effects (glutamate and glutamine) in macrophages. Taking together the above previous reports with the mechanisms behind macrophage foam cell formation and atherogenesis, it is possible that AAs could be anti-atherogenic or pro-atherogenic via their mechanism of action on macrophage foam cell formation. This paradigm may serve as a basis for the development of novel cardio-protective, anti-atherogenic nutritional, or therapeutic approaches, that should be studied in human trials.

DETAILED DESCRIPTION:
Atherosclerosis is the underlying cause of cardiovascular diseases (CVD), the major cause of death worldwide. Atherosclerosis is an inflammatory disease of the arteries in which activated macrophages are abundant in the atherosclerotic lesions. Macrophages play key roles during early atherogenesis. After differentiating from peripheral blood monocytes, the formed intimal macrophages take up oxidized/modified lipoproteins and are transformed into lipid-rich foam cells, the hallmark feature of early atherogenesis. In addition to lipoprotein uptake, lipid accumulation in macrophages can also result from alterations in cellular lipid metabolism, e.g. attenuated reverse lipid transport or enhanced rates of lipid biosynthesis. Although much progress has been made in understanding the role of different lipids (fatty acids, cholesterol, phospholipids or triglycerides) in macrophage foam-cell formation and atherosclerosis development, little is known about the potential impact of other nutrients, such as amino acids (AAs).

Previous studies have demonstrated an association between specific AAs and increased CVD risk or higher prevalence of coronary artery disease (CAD). For instance, the role of the branched chain AAs (BCAAs; valine, leucine, and isoleucine) in atherogenesis and CVD has been recently studied. Association studies showed that the plasma levels of BCAAs significantly and independently correlated with dyslipidemia and CAD. However, BCAAs were found to possess cardio-protective effects in a heart failure rat model. Specifically, leucine was reported to attenuate atherosclerosis development in the atherosclerotic apoE-deficient (apoE-/-) mice model, by improving the plasma lipid profile and by reducing systemic inflammation. Other studies have indicated the ability of some AAs to exert anti-atherogenic effects. Glycine, the simplest AA, was inversely associated with the risk of acute myocardial infarction (AMI) in patients with high apolipoprotein B (apoB) and LDL-cholesterol levels. Cysteine is an essential AA in the biosynthesis of glutathione, a key endogenous anti-oxidant known for its anti-atherogenic properties in macrophage lipid metabolism leading to the attenuation of atherosclerosis development. Cysteine analogues such as N-acetyl cysteine (NAC) or ribose cysteine were shown to be anti-atherogenic. Arginine, a basic AA, is the main precursor for nitric oxide production in the vascular endothelium. Arginine was shown to protect endothelial cells from lipid peroxidation, and to delay or reduce atheroma formation. Arginine anti-atherogenicity includes its anti-oxidant properties and its ability to improve endothelial function in CVD or overweight patients.

The aim of the proposed study is to investigate the effects of one month of supplementation with specific AAs on changes in the macrophage atherogenicity and lipid metabolism together with other risk markers of atherosclerosis development, such as serum oxidative status and lipid levels, on healthy subjects. Findings from the current proposed study may shed light on yet unknown mechanisms by which specific AAs affect atherosclerosis development and CVD risk and hence could possibly assist in the future development of anti-atherogenic strategies

ELIGIBILITY:
Inclusion Criteria:

* healthy adult males between the ages of 18-50 after signing informed consent

Exclusion Criteria:

* pregnancy, renal, pulmonary, cardiovascular or endocrinal diseases, diabetes, cancer, morbid obesity (body mass index, BMI > 40 kg/m2), heavy smoking (> 20 cigarettes/day), or consumption of more than two alcoholic drinks per day. Subjects from the same hospital unit or from the laboratory where this study is conducted are also excluded

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-12-15 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Serum atherogenicity | 1 year
  Macrophage lipids (triglycerides and cholesterol) content (μg/mg cell protein) following incubation with serum derived from the subjects.

SECONDARY OUTCOMES:
Serum triglyceride concentration | 1 year
  Triglyceride concentration (mg/dL) vs control group
Macrophage cholesterol content | 1 year
  Cholesterol concentration (mg/dL) vs control group
Serum oxidation | 1 year
  Serum levels of thiobarbituric acid reactive substances (TBARS)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Hayek, Prof, Principal Investigator — Rambam Health Care Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Michas G, Micha R, Zampelas A. Dietary fats and cardiovascular disease: putting together the pieces of a complicated puzzle. Atherosclerosis. 2014 Jun;234(2):320-8. doi: 10.1016/j.atherosclerosis.2014.03.013. Epub 2014 Mar 27. PMID 24727233
- [Background] Dickhout JG, Basseri S, Austin RC. Macrophage function and its impact on atherosclerotic lesion composition, progression, and stability: the good, the bad, and the ugly. Arterioscler Thromb Vasc Biol. 2008 Aug;28(8):1413-5. doi: 10.1161/ATVBAHA.108.169144. No abstract available. PMID 18650503
- [Background] Rom O, Aviram M. Endogenous or exogenous antioxidants vs. pro-oxidants in macrophage atherogenicity. Curr Opin Lipidol. 2016 Apr;27(2):204-6. doi: 10.1097/MOL.0000000000000287. No abstract available. PMID 26959710
- [Background] Afonso Mda S, Castilho G, Lavrador MS, Passarelli M, Nakandakare ER, Lottenberg SA, Lottenberg AM. The impact of dietary fatty acids on macrophage cholesterol homeostasis. J Nutr Biochem. 2014 Feb;25(2):95-103. doi: 10.1016/j.jnutbio.2013.10.001. Epub 2013 Oct 31. PMID 24445035
- [Background] Huang Y, Zhou M, Sun H, Wang Y. Branched-chain amino acid metabolism in heart disease: an epiphenomenon or a real culprit? Cardiovasc Res. 2011 May 1;90(2):220-3. doi: 10.1093/cvr/cvr070. PMID 21502372
- [Background] Yang RY, Wang SM, Sun L, Liu JM, Li HX, Sui XF, Wang M, Xiu HL, Wang S, He Q, Dong J, Chen WX. Association of branched-chain amino acids with coronary artery disease: A matched-pair case-control study. Nutr Metab Cardiovasc Dis. 2015 Oct;25(10):937-42. doi: 10.1016/j.numecd.2015.06.003. Epub 2015 Jun 14. PMID 26231617
- [Background] Shah SH, Bain JR, Muehlbauer MJ, Stevens RD, Crosslin DR, Haynes C, Dungan J, Newby LK, Hauser ER, Ginsburg GS, Newgard CB, Kraus WE. Association of a peripheral blood metabolic profile with coronary artery disease and risk of subsequent cardiovascular events. Circ Cardiovasc Genet. 2010 Apr;3(2):207-14. doi: 10.1161/CIRCGENETICS.109.852814. Epub 2010 Feb 19. PMID 20173117
- [Background] Bhattacharya S, Granger CB, Craig D, Haynes C, Bain J, Stevens RD, Hauser ER, Newgard CB, Kraus WE, Newby LK, Shah SH. Validation of the association between a branched chain amino acid metabolite profile and extremes of coronary artery disease in patients referred for cardiac catheterization. Atherosclerosis. 2014 Jan;232(1):191-6. doi: 10.1016/j.atherosclerosis.2013.10.036. Epub 2013 Nov 12. PMID 24401236
- [Background] Tanada Y, Shioi T, Kato T, Kawamoto A, Okuda J, Kimura T. Branched-chain amino acids ameliorate heart failure with cardiac cachexia in rats. Life Sci. 2015 Sep 15;137:20-7. doi: 10.1016/j.lfs.2015.06.021. Epub 2015 Jul 2. PMID 26141987
- [Background] Zhao Y, Dai XY, Zhou Z, Zhao GX, Wang X, Xu MJ. Leucine supplementation via drinking water reduces atherosclerotic lesions in apoE null mice. Acta Pharmacol Sin. 2016 Feb;37(2):196-203. doi: 10.1038/aps.2015.88. Epub 2015 Dec 21. PMID 26687933
- [Background] Wurtz P, Raiko JR, Magnussen CG, Soininen P, Kangas AJ, Tynkkynen T, Thomson R, Laatikainen R, Savolainen MJ, Laurikka J, Kuukasjarvi P, Tarkka M, Karhunen PJ, Jula A, Viikari JS, Kahonen M, Lehtimaki T, Juonala M, Ala-Korpela M, Raitakari OT. High-throughput quantification of circulating metabolites improves prediction of subclinical atherosclerosis. Eur Heart J. 2012 Sep;33(18):2307-16. doi: 10.1093/eurheartj/ehs020. Epub 2012 Mar 26. PMID 22450427
- [Background] Selhub J, Troen AM. Sulfur amino acids and atherosclerosis: a role for excess dietary methionine. Ann N Y Acad Sci. 2016 Jan;1363:18-25. doi: 10.1111/nyas.12962. Epub 2015 Dec 8. PMID 26647293
- [Background] Toborek M, Kopieczna-Grzebieniak E, Drozdz M, Wieczorek M. Increased lipid peroxidation as a mechanism of methionine-induced atherosclerosis in rabbits. Atherosclerosis. 1995 Jun;115(2):217-24. doi: 10.1016/0021-9150(94)05516-l. PMID 7661880
- [Background] Julve J, Escola-Gil JC, Rodriguez-Millan E, Martin-Campos JM, Jauhiainen M, Quesada H, Renteria-Obregon IM, Osada J, Sanchez-Quesada JL, Blanco-Vaca F. Methionine-induced hyperhomocysteinemia impairs the antioxidant ability of high-density lipoproteins without reducing in vivo macrophage-specific reverse cholesterol transport. Mol Nutr Food Res. 2013 Oct;57(10):1814-24. doi: 10.1002/mnfr.201300133. Epub 2013 Jun 10. PMID 23754667
- [Background] Yang AN, Zhang HP, Sun Y, Yang XL, Wang N, Zhu G, Zhang H, Xu H, Ma SC, Zhang Y, Li GZ, Jia YX, Cao J, Jiang YD. High-methionine diets accelerate atherosclerosis by HHcy-mediated FABP4 gene demethylation pathway via DNMT1 in ApoE(-/-) mice. FEBS Lett. 2015 Dec 21;589(24 Pt B):3998-4009. doi: 10.1016/j.febslet.2015.11.010. Epub 2015 Nov 26. PMID 26606905
- [Background] Ding Y, Svingen GF, Pedersen ER, Gregory JF, Ueland PM, Tell GS, Nygard OK. Plasma Glycine and Risk of Acute Myocardial Infarction in Patients With Suspected Stable Angina Pectoris. J Am Heart Assoc. 2015 Dec 31;5(1):e002621. doi: 10.1161/JAHA.115.002621. PMID 26722126
- [Background] Rosenblat M, Volkova N, Coleman R, Aviram M. Anti-oxidant and anti-atherogenic properties of liposomal glutathione: studies in vitro, and in the atherosclerotic apolipoprotein E-deficient mice. Atherosclerosis. 2007 Dec;195(2):e61-8. doi: 10.1016/j.atherosclerosis.2007.05.012. Epub 2007 Jun 22. PMID 17588583
- [Background] Kader T, Porteous CM, Williams MJ, Gieseg SP, McCormick SP. Ribose-cysteine increases glutathione-based antioxidant status and reduces LDL in human lipoprotein(a) mice. Atherosclerosis. 2014 Dec;237(2):725-33. doi: 10.1016/j.atherosclerosis.2014.10.101. Epub 2014 Nov 1. PMID 25463112
- [Background] Suschek CV, Schnorr O, Hemmrich K, Aust O, Klotz LO, Sies H, Kolb-Bachofen V. Critical role of L-arginine in endothelial cell survival during oxidative stress. Circulation. 2003 May 27;107(20):2607-14. doi: 10.1161/01.CIR.0000066909.13953.F1. Epub 2003 May 12. PMID 12742995
- [Background] Wang BY, Ho HK, Lin PS, Schwarzacher SP, Pollman MJ, Gibbons GH, Tsao PS, Cooke JP. Regression of atherosclerosis: role of nitric oxide and apoptosis. Circulation. 1999 Mar 9;99(9):1236-41. doi: 10.1161/01.cir.99.9.1236. PMID 10069793
- [Background] Deveaux A, Pham I, West SG, Andre E, Lantoine-Adam F, Bunouf P, Sadi S, Hermier D, Mathe V, Fouillet H, Huneau JF, Benamouzig R, Mariotti F. l-Arginine Supplementation Alleviates Postprandial Endothelial Dysfunction When Baseline Fasting Plasma Arginine Concentration Is Low: A Randomized Controlled Trial in Healthy Overweight Adults with Cardiometabolic Risk Factors. J Nutr. 2016 Jul;146(7):1330-40. doi: 10.3945/jn.115.227959. Epub 2016 Jun 8. PMID 27281800
- [Background] Rom O, Grajeda-Iglesias C, Najjar M, Abu-Saleh N, Volkova N, Dar DE, Hayek T, Aviram M. Atherogenicity of amino acids in the lipid-laden macrophage model system in vitro and in atherosclerotic mice: a key role for triglyceride metabolism. J Nutr Biochem. 2017 Jul;45:24-38. doi: 10.1016/j.jnutbio.2017.02.023. Epub 2017 Apr 6. PMID 28431321
- [Background] Eierman DF, Johnson CE, Haskill JS. Human monocyte inflammatory mediator gene expression is selectively regulated by adherence substrates. J Immunol. 1989 Mar 15;142(6):1970-6. PMID 2784145
- [Result] Nikitina NA, Sobenin IA, Myasoedova VA, Korennaya VV, Mel'nichenko AA, Khalilov EM, Orekhov AN. Antiatherogenic effect of grape flavonoids in an ex vivo model. Bull Exp Biol Med. 2006 Jun;141(6):712-5. doi: 10.1007/s10517-006-0260-7. English, Russian. PMID 17364057
- [Result] Hamoud S, Hayek T, Volkova N, Attias J, Moscoviz D, Rosenblat M, Aviram M. Pomegranate extract (POMx) decreases the atherogenicity of serum and of human monocyte-derived macrophages (HMDM) in simvastatin-treated hypercholesterolemic patients: a double-blinded, placebo-controlled, randomized, prospective pilot study. Atherosclerosis. 2014 Jan;232(1):204-10. doi: 10.1016/j.atherosclerosis.2013.11.037. Epub 2013 Nov 19. PMID 24401239
- [Result] Trumbo P, Schlicker S, Yates AA, Poos M; Food and Nutrition Board of the Institute of Medicine, The National Academies. Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids. J Am Diet Assoc. 2002 Nov;102(11):1621-30. doi: 10.1016/s0002-8223(02)90346-9. No abstract available. PMID 12449285